CLINICAL TRIAL: NCT03303534
Title: Short-Term Endogenous Hydrogen Sulfide Upregulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, C. Keith Ozaki, M.D., F.A.C.S., Attending Surgeon, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2016P002507
Record Dates: First submitted 2017-09-27; First posted 2017-10-06 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Carotid Stenosis; Caloric Restriction
Keywords: inflammation; hydrogen sulfide; caloric restriction; vascular surgery
MeSH Terms: conditions — Carotid Stenosis; Inflammation

STUDY DESIGN:
Intervention Model Description: 3:2 randomization to short-term protein calorie restriction diet versus regular meals prior to elective carotid artery endarterectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCR (Experimental): pre-operative protein calorie restricted (PCR) group. participants randomized to this arm will consume scandishake diet (strawberry, caramel, banana cream, vanilla) mixed with almond milk for three days inpatient prior to planned elective carotid endarterectomy. Water is ad libitum for this cohort. Nutritionists will prepare shakes so participants will achieve 30% calorie restriction and severe protein restriction during the three days on the diet.
  Interventions: Dietary Supplement: ScandiShake
- control regular diet (No Intervention): participants in this cohort are randomized to the control group and will have no dietary restriction three days in patient prior to planned elective carotid endarterectomy

INTERVENTIONS:
Dietary Supplement: ScandiShake — weight gain supplement low in protein
  Arms: PCR

SUMMARY:
This research study will compare the impact of dietary restriction pre-operatively before carotid endarterectomy compared to the standard nutrition that a patient typically eats. The investigators want to find out how patients comply and generally how well patients do with this type of dietary restriction before their surgery since animal studies suggest that short - term dietary restriction may be beneficial before surgery.

DETAILED DESCRIPTION:
The primary, scientific long term objective is to study any correlation that brief upregulation of endogenous hydrogen sulfide (H2S) via pre-operative protein calorie restriction (PCR) in elective major surgery may have biologic effects in humans. In this study, the investigators plan to evaluate patient compliance and the physiologic response pre-operative PCR has on patients undergoing carotid endarterectomy surgery. This will be explored via two primary aims.

The First Aim looks to create a prospective, fast-track, one-year study of 40 vascular surgery patients undergoing elective carotid artery endarterectomy randomized into two pre-operative dietary groups: observational group (n=16) and PCR (commercially available ScandiShake x 3 days, n=24). This pilot study is based on preliminary data balanced with economic and clinical feasibility considerations. The primary endpoints of this study are: 1) feasibility of subject compliance with PCR (measured by direct dietary intake data and serum markers including plasma free amino acids and insulin-like growth factor; thus the 2:3 randomization) and 2) measurement of H2S and standard markers of stress before and after surgery (including stress hormones, oxidative stress, inflammation and cardiac troponin T levels). Individual patient's microbiomes,phenotype of circulating blood cells, adipose tissue (peri-vascular, subcutaneous), and the excised carotid plaque will be characterized to inform on potential mechanistic links among these and PCR induced H2S upregulation, reduced peri-operative stress, atherosclerotic plaque stability, and improved outcome (baseline and peri-procedural clinical datasets will be completed) for future clinical trials. Key secondary data points include observing endpoints such as carotid restenosis and surgical complications (cardiac, neurologic, wound, etc) between the two groups, which the investigators hypothesize will help to inform future trials. This pilot study will elucidate not only the practicality of pre-operative short term dietary restriction, but also provide physiologic data to support the long term primary scientific objective stated previously.

The Second Specific Aim is to establish a robust human discovery multi-institutional platform to capitalize on multiple aspects of this carefully constructed initiative toward long-term goals such as better understanding and translation of the biologic mechanisms of H2S and PCR. Data collected in the first aim across institutions will be integrated and made public.This platform will encourage communication and collaboration among basic scientists, translational investigators, and clinical communities. This synergy will allow the investigators to define the mechanisms of H2S and PCR effects, and will also give insights into the human response to trauma (lipidomics, microbiome, proteins/microRNAs) that regulate the pro-inflammatory response to injury, and will allow for mechanistic links among these factors ties to surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* consenting adults (men and women)
* clinical indication for carotid endarterectomy (CEA) as determined by attending vascular surgeon
* if symptomatic, patients must be able to safely have surgery timed for PCR intervention

Exclusion Criteria:

* intolerance or allergy to any ingredients in the PCR diet (ScandiShake ingredients or almond milk/nuts)
* active infection
* pregnancy
* malnutrition determined by serum albumin lower than BWH reference value of 3.5 g/dL
* active drug dependency or alcoholism that could interfere with protocol adherence
* active non-cutaneous cancer under treatment with chemotherapeutic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
subject compliance with PCR | three days pre-operatively
  will measure subject compliance via direct dietary intake data by way of written food diary and biologic markers (serum markers including plasma free amino acids and insulin-like growth factor).

SECONDARY OUTCOMES:
measurement of local and systemic hydrogen sulfide and standard markers of stress peri-procedurally | change over 4.5 weeks from baseline
  hydrogen sulfide upregulation has been linked to improved vascular surgery outcomes in rodent models when rodents are pre-operatively on PCR diets
fecal microbiome characterization | change over 4.5 weeks from baseline
  if PCR and surgery has an impact on patient microbiome or microbiome related metabolites

CONTACTS AND LOCATIONS:
Overall Officials: C. Keith Ozaki, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hine C, Kim HJ, Zhu Y, Harputlugil E, Longchamp A, Matos MS, Ramadoss P, Bauerle K, Brace L, Asara JM, Ozaki CK, Cheng SY, Singha S, Ahn KH, Kimmelman A, Fisher FM, Pissios P, Withers DJ, Selman C, Wang R, Yen K, Longo VD, Cohen P, Bartke A, Kopchick JJ, Miller R, Hollenberg AN, Mitchell JR. Hypothalamic-Pituitary Axis Regulates Hydrogen Sulfide Production. Cell Metab. 2017 Jun 6;25(6):1320-1333.e5. doi: 10.1016/j.cmet.2017.05.003. PMID 28591635
- [Background] Longchamp A, Harputlugil E, Corpataux JM, Ozaki CK, Mitchell JR. Is Overnight Fasting before Surgery Too Much or Not Enough? How Basic Aging Research Can Guide Preoperative Nutritional Recommendations to Improve Surgical Outcomes: A Mini-Review. Gerontology. 2017;63(3):228-237. doi: 10.1159/000453109. Epub 2017 Jan 5. PMID 28052287
- [Background] Longchamp A, Tao M, Bartelt A, Ding K, Lynch L, Hine C, Corpataux JM, Kristal BS, Mitchell JR, Ozaki CK. Surgical injury induces local and distant adipose tissue browning. Adipocyte. 2015 Nov 20;5(2):163-74. doi: 10.1080/21623945.2015.1111971. eCollection 2016 Apr-Jun. PMID 27386152
- [Background] Robertson LT, Trevino-Villarreal JH, Mejia P, Grondin Y, Harputlugil E, Hine C, Vargas D, Zheng H, Ozaki CK, Kristal BS, Simpson SJ, Mitchell JR. Protein and Calorie Restriction Contribute Additively to Protection from Renal Ischemia Reperfusion Injury Partly via Leptin Reduction in Male Mice. J Nutr. 2015 Aug;145(8):1717-27. doi: 10.3945/jn.114.199380. Epub 2015 Jun 3. PMID 26041674
- [Background] Hine C, Harputlugil E, Zhang Y, Ruckenstuhl C, Lee BC, Brace L, Longchamp A, Trevino-Villarreal JH, Mejia P, Ozaki CK, Wang R, Gladyshev VN, Madeo F, Mair WB, Mitchell JR. Endogenous hydrogen sulfide production is essential for dietary restriction benefits. Cell. 2015 Jan 15;160(1-2):132-44. doi: 10.1016/j.cell.2014.11.048. Epub 2014 Dec 23. PMID 25542313
- [Background] Mauro CR, Tao M, Yu P, Trevino-Villerreal JH, Longchamp A, Kristal BS, Ozaki CK, Mitchell JR. Preoperative dietary restriction reduces intimal hyperplasia and protects from ischemia-reperfusion injury. J Vasc Surg. 2016 Feb;63(2):500-9.e1. doi: 10.1016/j.jvs.2014.07.004. Epub 2014 Aug 8. PMID 25124359
- [Background] Nguyen B, Tao M, Yu P, Mauro C, Seidman MA, Wang YE, Mitchell J, Ozaki CK. Preoperative diet impacts the adipose tissue response to surgical trauma. Surgery. 2013 Apr;153(4):584-93. doi: 10.1016/j.surg.2012.11.001. Epub 2012 Dec 27. PMID 23274098
- [Background] Mitchell JR, Beckman JA, Nguyen LL, Ozaki CK. Reducing elective vascular surgery perioperative risk with brief preoperative dietary restriction. Surgery. 2013 Apr;153(4):594-8. doi: 10.1016/j.surg.2012.09.007. Epub 2012 Dec 4. PMID 23218877